CLINICAL TRIAL: NCT06570161
Title: Assessment of User Preference and Fit of Novel Transparent Face Masks
Brief Title: Assessment of Fit of Novel N95 Style Transparent Face Masks
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: funding terminated
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Peter R Chai MD, Associate Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2024P001913
Record Dates: First submitted 2024-08-15; First posted 2024-08-26 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Respiratory Disease; Infection, Coronavirus; Respiratory Tract Infections
MeSH Terms: conditions — Respiration Disorders; Coronavirus Infections; Respiratory Tract Infections | interventions — N95 Respirators

STUDY DESIGN:
Intervention Model Description: Randomized crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SEEUS95 (Experimental): Transparent mask developed by SEEUS95
  Interventions: Device: SEEUS95 Transparent mask
- CrystalGuard (Experimental): Transparent mask developed at BWH
  Interventions: Device: CrystalGuard Mask
- N95 (Active Comparator): Standard N95 face mask
  Interventions: Device: N95 face mask

INTERVENTIONS:
Device: SEEUS95 Transparent mask — SEEUS95 developed transparent filtering mask
  Other Names: SEEUS95
  Arms: SEEUS95
Device: CrystalGuard Mask — CrystalGuard transparent mask
  Other Names: CrystalGuard
  Arms: CrystalGuard
Device: N95 face mask — Standard N95 style face mask
  Other Names: N95
  Arms: N95

SUMMARY:
Face masks have become a critically important public health intervention after the COVID-19 pandemic. Multiple types of masks ranging from full face filtering to cloth masks have been developed and commercialized to facilitate protection against respiratory pathogens. Most of these systems are made with opaque fabrics and may prevent individuals from expressing emotions or for those who are deaf and hard of hearing, communicating. To date, few transparent face masks which also confer respiratory pathogen protection have been developed. This study will test the feasability and acceptability of two new masks, the SEEUS-95 mask and CrystalGuard mask which are both transparent versions of N-95 filtering face masks.

DETAILED DESCRIPTION:
This is a randomized crossover trial to evaluate the feasibility, acceptability and choice between the use of the SEEUS-95, CrystalGuard transparent face masks or a standard N95 mask. Otherwise healthy individuals will be prescreened and then scheduled for a single study visit. Participants will be randomized to wear each of the three masks (SEEUS-95, CrystalGuard, N95). They will be taught how to wear the mask, and we will assist participants with correctly wearing the mask for a good fit. Next, participants will undergo standard FIT testing where a clear hood will be placed over the participant's head, and a bitter solution (Bitrex) is sprayed into the hood. A positive test is indicated if the participant is able to taste Bitrex demonstrating that there is a detected leak within the mask. After a few minute washout period, participants will undergo FIT testing of subsequent masks. We will ask participants to rate the comfort of wearing the masks, willingness to wear masks in public and suggestions for improvement in mask design. Finally, we will conduct a discrete choice test to ask participants which mask they would prefer to wear in public.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* No history of asthma, restrictive lung disease, interstitial lung disease, or emphysema
* Lack of significant facial hair that precludes wearing a N-95 mask

Exclusion Criteria:

* Less than 18 years old
* Unable to smell Bitrex solution used for fit testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability | immediately after mask wearing
  User acceptability and comfort wearing the assigned mask graded on a likert scale

SECONDARY OUTCOMES:
Mask preference | immediately after completion of all three arms
  Discrete choice of SEEUS-95, CrystalGuard versus standard N-95 mask selected by study participants

CONTACTS AND LOCATIONS:
Overall Officials: Peter Chai, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No